CLINICAL TRIAL: NCT02329938
Title: Desarda Versus Lichtenstein's Repair for Inguinal Hernia: a Comparative Study
Brief Title: Desarda Repair for Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tamer Youssef Mohamed, assistant professor of surgery, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MFM200956
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Lichtenstein tension free reair (Active Comparator): mesh repair of inguinal hernia
  Interventions: Procedure: Lichtenstein tension free reair
- Desarda's repair (Active Comparator): non-mesh repair of inguinal hernia
  Interventions: Procedure: Desarda's repair

INTERVENTIONS:
Procedure: Lichtenstein tension free reair — a mesh is apllied on the posterior wall of the inguinal canal and sutured to the inguinal ligament below, to the internal oblique muscle above , and to rectus sheath medially.
  Other Names: pure synthetic repair
  Arms: Lichtenstein tension free reair
Procedure: Desarda's repair — the repair is done using a flap of the external oblique aponeurosis sutured to the inguinal ligament below and to the aponeurotic part of the internal oblique muscle above.
  Other Names: pure tissue reapir
  Arms: Desarda's repair

SUMMARY:
Unlike Lichtenstein tension free repair for inguinal hernia, Desarda's repair was introduced as a pure tissue repair with no need for mesh. In other words; the complications which may arise from the use of a foreign body (mesh) will be avoided. The idea was to evaluate the efficacy of this new repair and compare it to the standard Lichtenstein repair.

ELIGIBILITY:
Inclusion Criteria:

* inguinal hernia

Exclusion Criteria:

* recurrent inguinal hernia
* giant inguinal hernia
* mental disorder
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
number of patients with recurrence of inguinal hernia | 2 years

SECONDARY OUTCOMES:
VAS score for pain | one year
number of patients develped postoperative complications | 2 years

REFERENCES:
- [Derived] Youssef T, El-Alfy K, Farid M. Randomized clinical trial of Desarda versus Lichtenstein repair for treatment of primary inguinal hernia. Int J Surg. 2015 Aug;20:28-34. doi: 10.1016/j.ijsu.2015.05.055. Epub 2015 Jun 11. PMID 26074293